CLINICAL TRIAL: NCT04809558
Title: Determining an Optimal Delivery Method for Tongue Strengthening During Swallowing Rehabilitation: Building a Framework for Clinical Practice
Brief Title: Optimal Method for Tongue Strengthening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samford University (Other)
Collaborators: Case Western Reserve University (Other); Emerson College (Other); James Madison University (Other); Texas Christian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXPD-HP-20-F-5
Record Dates: First submitted 2021-03-12; First posted 2021-03-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2022-12

CONDITIONS: Focus of Study is Tongue Strength

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will only know exercise instructions for the group he/she is randomized to. Participant will not be provided with information about other groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Max intensity with no visual biofeedback (Active Comparator): Tongue resistance exercises completed at maximum intensity with no visual biofeedback.
  Interventions: Behavioral: Tongue resistance exercise
- Progressive intensity with no visual biofeedback. (Active Comparator): Tongue resistance exercises completed at a progressive intensity with no visual biofeedback.
  Interventions: Behavioral: Tongue resistance exercise
- Max intensity with visual biofeedback (Active Comparator): Tongue resistance exercises completed at maximum intensity with visual biofeedback of performance.
  Interventions: Behavioral: Tongue resistance exercise
- Progressive intensity with visual biofeedback. (Active Comparator): Tongue resistance exercises completed at a progressive intensity with visual biofeedback of performance.
  Interventions: Behavioral: Tongue resistance exercise

INTERVENTIONS:
Behavioral: Tongue resistance exercise — Participant will complete tongue resistance exercises.

SUMMARY:
The research team will conduct a multi-site, randomized controlled trial examining the effectiveness of exercise intensity progression compared to standard practice (no progression) in the context of swallowing rehabilitation. The study will also determine the impact of using biofeedback during resistance training on tongue strength. The study is a first step in determining an optimal delivery of tongue strengthening exercise in typically aging older persons, with the plan to develop a framework for guiding clinical practice of tongue strengthening in various dysphagic populations. Participants will be randomized into one of four treatment groups and complete 8 weeks of tongue resistance training.

DETAILED DESCRIPTION:
Rehabilitative exercises have been central to dysphagia (swallowing difficulty) treatment for decades, with the goal to increase strength, endurance, and/or coordination of the muscles responsible for swallowing. With any exercise-based therapy, an understanding of dosing is critical to optimize outcomes and to avoid over- or under-prescribing exercise, which can have a negative effect. For example, overtraining can lead to reductions in strength, which may put patients who are completing a swallowing rehabilitation program at increased risk. Therefore, it is important to develop dosing recommendations specific to swallowing musculature. Clinical practice remains unguided in terms of whether a progressive or maximum intensity, both common forms of rehabilitative exercise for dysphagic patients, should be used for lingual resistance training. Speech-Language Pathologists (SLP) currently base these decisions on preference and experience; however, research is desperately needed in this area to support and guide clinical decisions. The investigators aim to fill this gap in evidence by determining an optimal dosing for tongue strengthening in older persons. It is anticipated that the study findings will directly influence clinical decisions in both inpatient rehabilitation facilities and home health post-acute care settings, and ultimately improve patient outcomes in the area of swallowing. This study represents the start of a research program intended to provide significant information on optimal delivery of tongue strengthening exercise in various populations with difficulty swallowing.

To determine an optimal delivery method for tongue resistance training in healthy older persons by examining how intensity progression and biofeedback impacts tongue strength, participant motivation, and program adherence. The data collected in this initial study will inform future studies designed to develop a framework for guiding clinical practice with SLPs prescribing tongue strengthening exercise to patients with swallowing issues.

Primary Research Questions:

* Is tongue strength impacted by exercise resistance intensity when comparing progressive resistance to maximum resistance?
* Is tongue strength impacted by visual biofeedback during tongue resistance training?

Secondary Research Questions:

* Is participant motivation impacted by progressive intensity exercise when compared to maximum intensity exercise?
* Is participant motivation impacted by the use of biofeedback when compared to no visual biofeedback?
* Is participant adherence to the exercise program impacted by progressive intensity exercise when compared to maximum intensity exercise?
* Is participant adherence to the exercise program impacted by the use of biofeedback when compared to no visual biofeedback?

ELIGIBILITY:
Inclusion Criteria:

* Are age 55 or older
* < 3 score on Eating Assessment Tool-10 (screening tool for swallowing difficulty)
* > 24 score on Mini Mental State Examination (screening tool for cognitive impairment)
* Have a normal oral structure as assessed with an oral mechanism screener

Exclusion Criteria:

* A history of seizures (contraindication for Tongueometer™ use)
* Past or present pain disorders involving the jaw or mandible (e.g., TMJ disorder, myofascial pain disorder) (contraindication for Tongueometer™ use)
* A history of oral surgery (routine dental surgery acceptable)
* A history of neurogenic disorder (e.g., Parkinson's disease)
* A history of swallowing difficulty
* Not being able to complete an 8-week study protocol

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Change in maximum isometric tongue pressure (MIP) | Multiple baselines (2), every 2 weeks following for 8 weeks, 1-month post if person randomized to a maintenance program
  MIP in kilopascals (kPa)
Change in regular effort saliva swallow pressure (RESS) | Multiple baselines (2), every 2 weeks following for 8 weeks, 1-month post if person randomized to a maintenance program
  RESS is kilopascals (kPa)
Change in effortful swallow pressure (ESP) | Multiple baselines (2), every 2 weeks following for 8 weeks, 1-month post if person randomized to a maintenance program
  ESP in kilopascals (kPa)

SECONDARY OUTCOMES:
Change in participant-perceived motivation for assigned exercise regimen | Multiple baselines (2), every 2 weeks following for 8 weeks, 1-month post if person randomized to a maintenance program
  Standardized 0 mm (lowest level of perceived motivation) to 100 mm (highest level of perceived motivation) visual-analog scale participant perception of internal motivation.
Change in participant-perceived confidence for assigned exercise regimen | Multiple baselines (2), every 2 weeks following for 8 weeks, 1-month post if person randomized to a maintenance program
  Standardized 0 mm (lowest level of perceived confidence) to 100 mm (highest level of perceived confidence) visual-analog scale participant perception of internal confidence.
Exercise adherence tracking | Collected at Weeks, 2, 4, 6, 8; and 1-month post if participant was randomized to a maintenance program
  Adherence tracking will be completed by asking participants to keep record form logs of sessions completed

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H Szynkiewicz, Ph.D., Principal Investigator — Samford University; Erin Kamarunas, Ph.D., Principal Investigator — James Madison University; Teresa Drulia, Ph.D., Principal Investigator — Texas Christian University; Lindsay Griffin, Ph.D., Principal Investigator — Emerson College; Rachel Mulheren, Ph.D., Principal Investigator — Case Western Reserve University
Locations (1):
- Samford University, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhea MR, Alvar BA, Burkett LN, Ball SD. A meta-analysis to determine the dose response for strength development. Med Sci Sports Exerc. 2003 Mar;35(3):456-64. doi: 10.1249/01.MSS.0000053727.63505.D4. PMID 12618576
- [Derived] Kamarunas E, Murray K, Drulia T, Szynkiewicz S, Griffin L, Mulheren R. Biofeedback and Exercise Load Affect Accuracy of Tongue Strength Exercise Performance. Dysphagia. 2025 Apr;40(2):489-500. doi: 10.1007/s00455-024-10751-w. Epub 2024 Aug 18. PMID 39154305